CLINICAL TRIAL: NCT05392465
Title: Effects of Holistic Spinal Fascial Mobilization on Pain, Range of Motion and Function in Patients With Chronic Neck Pain
Brief Title: Effects of Holistic Spinal Fascial Mobilization in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0144 Nimra
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
Keywords: Fascia; Range of motion; Mobilization
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): baseline physical therapy treatment along with facial mobilization
  Interventions: Other: Fascial mobilization group
- Group B (Other): baseline (Conventional) physical therapy treatment
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Fascial mobilization group — Fascial mobilization+ conventional treatment (3 sessions per week). MFR is thought to work directly on restricted fascia; practitioners use knuckles or elbow to slowly sink into the fascia, and the pressure applied to contact the restricted fascia, apply tension, or stretch the fascia. MFR involves application of gentle stretch the pressure applied is a few grams of force, and the hands tend to follow the direction of fascial restriction, hold the stretch, and allow the fascia to release itself + hot pack (10 min) + neck isometrics (neck flexion, extension, side bending) + neck stretches (neck flexors, extensors, side benders and rotation).A total of 40-45 min session three times a week on alternate days for three weeks.
  Arms: Group A
Other: Conventional physical therapy — Conventional Therapy (3 sessions per week). In this treatment group conventional treatment for chronic neck pain will be given which includes hot pack, Neck Isometrics and Neck Stretches. Hot pack (10 min) + neck isometrics (neck flexion, extension, side bending) + neck stretches (neck flexors, extensors, side benders and rotators).A total of 40-45 min session three times a week on alternate days for three weeks On eligible participants baseline assessment was done,3 session were given per week.
  Arms: Group B

SUMMARY:
This study aims to determine the effects of holistic spinal fascial mobilization on pain, range of motion and function in patients with chronic neck pain so that we can have the best treatment option for patients with chronic neck pain, the duration will be 10 months, purposive sampling will be done, subject following eligibility criteria from bahawal Victoria hospital Bahawalpur, were allocated in two groups, a baseline assessment was done, Group A participants were given conventional treatment along with fascial mobilization, Group B participants were given conventional treatment, Numeric pain rating scale(NPRS), Neck Disability Index(NDI) and Goniometry for a range of motion,3 sessions per week were given, data was analyzed by using SPSS version 25.

DETAILED DESCRIPTION:
Chronic neck pain is one of the most common musculoskeletal disorders among the general population. Like a muscular spasm of the neck that can cause neck pain, fascial adhesions are also a common cause of neck pain. Fascia is a form of connective tissue that is made up of collagen, surrounds the body parts, and also resists tissue tensile load. There is huge literature regarding the management of neck pain and yet after decades of research, there are gaps in treatment options. In the modern age of health care, it is a common goal of every health care to make patients self-sufficient as early as possible. The self-care models have tremendous advantages. The current study aims to determine the effects of holistic spinal fascial mobilization on pain, range of motion, and function in patients with chronic neck pain. All treatment methods were employed to see if they improve the ranges accompanying pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age 25-60 years.
* NPRS >4
* Subjects diagnosed with chronic neck pain with minimum 3 months of chronicity
* Subjects without any other pathology affecting the neck and upper limb.

Exclusion Criteria:

* Subjects with a history of Vertebro-Basilar artery insufficiency
* Any bony, soft tissue, systemic disease, fever, malnutrition or tumor.
* Surgery

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. Where 0 indicate no pain and 10 indicate severe pain
NDI | 3rd day
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. The maximum score is 5.
Goniometric measurement of Neck ROM | 3rd day
  A goniometer is an instrument which measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Bhawal Victoria Hospital, Bhawalpur, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McLean SM, May S, Klaber-Moffett J, Sharp DM, Gardiner E. Risk factors for the onset of non-specific neck pain: a systematic review. J Epidemiol Community Health. 2010 Jul;64(7):565-72. doi: 10.1136/jech.2009.090720. Epub 2010 May 12. PMID 20466711
- [Background] Chiu TT, Hui-Chan CW, Chein G. A randomized clinical trial of TENS and exercise for patients with chronic neck pain. Clin Rehabil. 2005 Dec;19(8):850-60. doi: 10.1191/0269215505cr920oa. PMID 16323384
- [Background] Bakry HA. The effect of poor posture on the cervical range of motion in young subjects. Egyptian Journal of Physical Therapy. 2021;5(1):5-12.
- [Background] Benjamin M. The fascia of the limbs and back--a review. J Anat. 2009 Jan;214(1):1-18. doi: 10.1111/j.1469-7580.2008.01011.x. PMID 19166469
- [Background] Hrkal P. Fascia: The Tensional Network of the Human Body: The science and clinical applications in manual and movement therapy. Journal of the Canadian Chiropractic Association. 2015;59(4):417-8.
- [Background] Laimi K, Makila A, Barlund E, Katajapuu N, Oksanen A, Seikkula V, Karppinen J, Saltychev M. Effectiveness of myofascial release in treatment of chronic musculoskeletal pain: a systematic review. Clin Rehabil. 2018 Apr;32(4):440-450. doi: 10.1177/0269215517732820. Epub 2017 Sep 28. PMID 28956477
- [Background] Rodriguez-Huguet M, Rodriguez-Almagro D, Rodriguez-Huguet P, Martin-Valero R, Lomas-Vega R. Treatment of Neck Pain With Myofascial Therapies: A Single Blind Randomized Controlled Trial. J Manipulative Physiol Ther. 2020 Feb;43(2):160-170. doi: 10.1016/j.jmpt.2019.12.001. Epub 2020 Apr 18. PMID 32317109
- [Background] Courraud C, Bertrand I, Dupuis C. Assessment of the effects of DBM fasciatherapy on fascial system with elastography.
- [Background] Quere N, Noel E, Lieutaud A, d'Alessio P. Fasciatherapy combined with pulsology touch induces changes in blood turbulence potentially beneficial for vascular endothelium. J Bodyw Mov Ther. 2009 Jul;13(3):239-45. doi: 10.1016/j.jbmt.2008.06.012. Epub 2008 Aug 12. PMID 19524848
- [Background] Stecco C, Day JA. The fascial manipulation technique and its biomechanical model: a guide to the human fascial system. Int J Ther Massage Bodywork. 2010 Mar 17;3(1):38-40. doi: 10.3822/ijtmb.v3i1.78. No abstract available. PMID 21589701